CLINICAL TRIAL: NCT04026490
Title: Evaluation of Link for Equity: A Program to Reduce Racial/Ethnic School Violence Disparities (Students of Color Population)
Brief Title: Evaluation of Link for Equity (Students of Color Population)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ExemptLinkEquityStudent; 1R01MD013801-01 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): The student will have a conversation with an Interventionist.
  Interventions: Behavioral: Immediate Intervention
- Waitlist intervention (Active Comparator): These students will be approached for intervention for the months following the implementation of the immediate intervention group using the same procedures.
  Interventions: Behavioral: Waitlist Intervention

INTERVENTIONS:
Behavioral: Immediate Intervention — The Interventionist will use motivational interviewing skills, assess ethnic and racial microaggressions, and provide support, screen for posttraumatic stress, and, if appropriate, link student to advanced care. The student may meet with the Interventionist several times during the remainder of the school year. These meetings will be approximately 10-30 minutes in length and occur during the school day in a private location determined by the Interventionist. The student may be referred to additional resources as a result of the meetings. The meetings will be documented by the Interventionist using a case management system (in RedCap).
  Arms: Immediate intervention
Behavioral: Waitlist Intervention — In order to compare outcomes contemporaneously, students from waitlisted schools will be asked to complete baseline and follow-up surveys, which will be collected at approximately the same time as in the immediate intervention schools. The data will be captured for analysis at the end of the study. Students will complete intervention following the waitlist period.
  Arms: Waitlist intervention

SUMMARY:
The investigators propose to develop and evaluate Link for Equity, a trauma-informed system of care. Link, a system of support for ACE-affected children, is composed of universal school Trauma-Informed Care. Preventing Racism through Awareness and Action (PRAA) is a perspective-taking racism/discrimination prevention intervention for school staff that increases awareness of racism and how it impacts students and promotes empathy for students of color. Link for Equity will be translated to be culturally responsive for 12 secondary public schools in metropolitan and rural Minnesota with substantial racial/ethnic minority students and racial/ethnic disparities in school discipline and violence. Using a nested, rigorous, and ethically acceptable randomized waitlist control design, the investigators will implement and evaluate Link for Equity sequentially for two years in each school. The overall goal is to evaluate if Link for Equity can reduce school violence disparities.

DETAILED DESCRIPTION:
Significance of Research Question/Purpose: Youth violence is an emergent nationwide public health issue. Almost two-thirds of public schools across America report one or more violent incidents on their campus annually. In 2014, approximately 850,000 non-fatal victimizations occurred among 12-18 year-old students; this includes 486,400 assaults and serious violent victimizations. About 22% of children in the U.S. reported being bullied at school in 2011, and one in 10 students report being threatened or injured with a weapon on school property in the past year.

Racial/ethnic minority youth are at increased risk for school violence. African American, Latino, and American Indian youth report higher rates of in-school physical fighting, weapon carrying, and gang presence compared to white youth. The highest rates of severe violence are reported in urban high schools with high minority enrollment, and large samples and reviews indicate Black and Latino youth engage in more bullying than other racial groups.

Accumulation of adverse child experiences (ACEs), or childhood traumas such as abuse, neglect, household dysfunction, and racial discrimination, place children at high risk for violent behaviors. Multiple ACEs are more prevalent among American Indian (40%), Hispanic (31%) and black children (33%) compared with white children (21%). ACEs have acute and cumulative detrimental impacts on the physiological, cognitive, behavioral and psychological health of children, and children with increased ACEs are more likely to engage in violent behaviors at school.

For example, the Olweus Anti-bullying Program, which was shown to be effective in Norway yet ineffective among Washington's racial/ethnic minority students, is implemented widely. A number of gaps in addressing risks for youth violence remain. Many programs are limited to didactic instruction in the classroom, or solely target children with significant behavioral concerns. Systems-based approaches are the most promising sustainable models because they capitalize on infrastructures and services offered at school. This study will evaluate a systems-based model, Link for Equity. Link is combines Trauma-Informed Care (TIC) and psychological first aid in a culturally sensitive manner. Link for Equity offers cultural humility training that specifically targets racial/ethnic microaggressions to prevent racial discrimination in discipline referrals of racial and ethnic minority students.

The aims are to:

Aim 1: Adapt, implement, and measure the effect of Link for Equity on school violence disparities.

Aim 2: Measure the effect of Link for Equity on racial discrimination by teachers (2a), and assess if teachers' racial discrimination mediates the effect of Link for Equity on school violence (2b).

Aim 3: Explore connectedness and stress mechanisms through which Link for Equity impacts school violence disparities.

ELIGIBILITY:
Inclusion Criteria:

* The student study population is composed of students of color enrolled at participating schools

Exclusion Criteria:

* Children who do not identify as full/part Black/African American, Latino/Hispanic, or American Indian/Native

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 518 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Change in School-based Racial and Ethnic Microaggressions Scale (SbREMS) Score | baseline and 2 years
  This is a 14-item scale that measures microaggressions that communicate perceptions of academic inferiority, expectations of aggression, and stereotypical misrepresentations. Respondents are instructed to indicate the number of times that a microaggression occurred in the past month from 1 (never) to 3 (regularly). Sub-scales include Academic Inferiority Microaggressions, Expectations of Aggression Microaggressions, and Stereotypical Misrepresentations Microaggressions. Items are averaged to obtain total and sub-scale scores. Higher scores indicate greater perceived frequency of racial microaggressions. Change in SbREMS score from baseline to two years post will be evaluated.
Change in Bullying incidents | baseline and 2 years
  Bullying is defined in Minnesota's anti-bullying law as recurrent aggression between peers leading to a power imbalance. Bullying perpetration and victimization will be evaluated in students enrolled in this study through semiannual surveys. Bullying perpetration and victimization incidents will also be examined using office referral and disciplinary action data from school records. Self-reported bullying is collected in the school-wide population through the Minnesota Student Survey, and will also be examined. From the secondary school measures, we will use counts per students enrolled. From the MSS data, we will report the change in the percentage of students who report an incident (e.g., percent bullied).
Change in Physical assault | baseline and 2 years
  Perpetration and victimization of physical assault, defined as physical harm against or by another student, will be evaluated using office referral and disciplinary action data from school records. Self-reported bullying is collected in the school-wide population through the Minnesota Student Survey, and will also be examined. From the secondary school measures, we will use counts per students enrolled. From the MSS data, we will report the change in the percentage of students who report an incident (e.g., percent of physical assaults).
Change in Weapons carrying | baseline and 2 years
  Minnesota law defines a dangerous weapon as any firearm, whether loaded or unloaded, or any device designed as a weapon or through its use is capable of threatening or producing death or great bodily harm. Weapons carrying will be evaluated using office referral and disciplinary action data from school records. From the secondary school measures, we will use counts per students enrolled. From the MSS data, we will report the change in the percentage of students who report an incident.
Change in Fighting | baseline and 2 years
  Incidents of fighting will be will be evaluated using office referral and disciplinary action data from school records. From the secondary school measures, we will use counts per students enrolled. From the MSS data, we will report the change in the percentage of students who report an incident.
Change in Subjective Disciplinary Practices | baseline and 2 years
  Subjective disciplinary practices are referrals and actions that are issued based on a subjective decision of teachers, including verbal abuse, defiance, disrespect, and dress code violations. Subjective disciplinary practices will be evaluated using office referral and disciplinary action data from school records. From the secondary school measures, we will use counts per students enrolled. From the MSS data, we will report the change in the percentage of students who report an incident.

CONTACTS AND LOCATIONS:
Overall Officials: Marizen Ramirez, PhD, MPH, Principal Investigator — University of Minnesota; Andrew Ryan, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez MR, Ryan A, Harding AB, Renfro T, Church TR, Rosebush C, Trotter AG, Xiong BN, Gonzalez J, Woods-Jaeger B. Link for Equity, a community-engaged waitlist randomized controlled trial of a culturally responsive trauma-informed care program for BIPOC students: Design features and characteristics of baseline sample. Contemp Clin Trials. 2023 Mar;126:107090. doi: 10.1016/j.cct.2023.107090. Epub 2023 Jan 18. PMID 36681238